CLINICAL TRIAL: NCT02897063
Title: The Effects of Midodrine and Droxidopa on Splanchnic Capacitance in Autonomic Failure Aim 2 of RDCRN (Rare Diseases Clinical Research Network) Project 2
Brief Title: Effects of Midodrine and Droxidopa on Splanchnic Capacitance in Autonomic Failure
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 160255
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2024-12

CONDITIONS: Autonomic Failure; Pure Autonomic Failure; Multiple System Atrophy; Parkinson Disease; Orthostatic Hypotension
Keywords: midodrine; droxidopa; splanchnic circulation
MeSH Terms: conditions — Pure Autonomic Failure; Multiple System Atrophy; Parkinson Disease; Hypotension, Orthostatic | interventions — Droxidopa; Midodrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Droxidopa and Placebo (Experimental): Patients will be studied on two separate days, two days apart: one day with the active drug and one day with placebo. The order of the study days will be randomized. On each study day, patients will receive a single oral dose of either droxidopa 300 mg or placebo after the first tilt table test, followed two hours later by a single oral dose of placebo.
  Interventions: Drug: Droxidopa; Drug: Placebo
- Midodrine and Placebo (Experimental): Patients will be studied on two separate days, two days apart: one day with the active drug and one day with placebo. The order of the study days will be randomized. On each study day, patients will receive a single oral dose of placebo after the first tilt table test, followed two hours later by a single oral dose of either midodrine 10 mg or placebo.
  Interventions: Drug: Midodrine; Drug: Placebo

INTERVENTIONS:
Drug: Droxidopa — Single oral dose 300 mg
  Other Names: Northera
  Arms: Droxidopa and Placebo
Drug: Midodrine — Single oral dose 10 mg
  Arms: Midodrine and Placebo
Drug: Placebo — sugar pill

SUMMARY:
The purpose of this study is to learn more about the effects of midodrine and droxidopa, two medications used for the treatment of orthostatic hypotension (low blood pressure on standing), on the veins of the abdomen of patients with autonomic failure. The study will be conducted at Vanderbilt University Medical Center, and consists of 2 parts: a screening and 2 testing days. The total length of the study will be about 5 days. About 34 participants will be screened for the study.

DETAILED DESCRIPTION:
Patients with multiple system atrophy, pure autonomic failure or Parkinson disease, and orthostatic hypotension will be studied in a randomized, double-blind, 2-arm parallel design to compare the effects of droxidopa and midodrine on stoke volume during head up tilt. A total of 34 participants will be enrolled in the study (17 patients in each arm).

Screening Procedures: Potential participants will be screened in the Vanderbilt Autonomic Dysfunction Center (ADC). Medications affecting blood pressure, blood volume and the autonomic nervous system such as pressor medications, fludrocortisone and carbidopa will be withdrawn for at least 5 half-lives before studies. Patients will undergo a complete history and physical examination, ECG, routine clinical laboratory analyses and a blood pregnancy test for women with childbearing potential. Autonomic testing including a tilt table testing and a posture study with plasma catecholamines is then performed to determine if they meet the inclusion/exclusion criteria.

Eligible participants will then be randomized to the droxidopa or the midodrine treatment group. All patients will be studied on two separate days, two days apart: one day with the active drug (droxidopa 300mg PO or midodrine 10mg PO) and one day with placebo.

On each study day, two tilt table tests will be performed. Patients will be instrumented to measure blood pressure and heart rate (continuously and intermittently), segmental impedance, cardiac output (inert gas rebreathing technique and/or impedance cardiography), and venous capacitance. Baseline measurements will then be taken in the supine position for about 30 minutes, and during head-up tilt for ≤10 minutes at 60 degrees. Supine baseline measurements will include the estimation of splanchnic venous capacitance. At the end of the head up tilt (HUT), patients will be asked to rate severity of their orthostatic symptoms.

Patients will then be placed in the seated position (time 0) and will receive a single oral dose of either droxidopa 300 mg or placebo, followed two hours later by a single oral dose of placebo or midodrine 10 mg. On the placebo day, both groups will receive a placebo pill at time 0 and at 2 hours. After ~3 hours of first drug administration, a second tilt table test will be performed, and outcome measurements will be repeated while supine and during HUT. The investigators may apply abdominal compression of 40 mmHg with an inflatable binder at the end of the second HUT. Outcome measurements will be repeated during 5 minutes of compression.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 40-80 years with possible or probable Multiple System Atrophy, Pure Autonomic Failure, or Parkinson disease, as defined by Consensus Criteria.
* Neurogenic orthostatic hypotension defined as a ≥30-mmHg decrease in systolic blood pressure within 3 minutes of standing associated with impaired autonomic reflexes determined by autonomic testing in the absence of other identifiable causes.
* Subjects able and willing to provide informed consent.

Exclusion Criteria:

* Supine hypertension, defined as systolic blood pressure of ≥ 160 mmHg measured on two separate occasions.
* Pregnancy.
* Systemic illnesses known to produce autonomic neuropathy, including but not limited to diabetes mellitus, amyloidosis, monoclonal gammopathies, and autoimmune neuropathies.
* History of known aortic aneurisms, thoracic, abdominal or pelvic surgery in the past 6 months.
* Symptomatic abdominal or inguinal hernias.
* Severe gastroesophageal reflux.
* Recent fractures or fissures of ribs, thoracic or lumbar spine.
* Medical devices implanted on the abdominal wall or abdomen that would interfere with the abdominal compression.
* Intolerance to any increase in intraabdominal pressure.
* Clinically unstable coronary artery disease or major cardiovascular or neurological event in the past 6 months, and other factors which in the investigator's opinion would prevent the subject from completing the protocol including clinically significant abnormalities in clinical, mental or laboratory testing.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-09; Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Stroke volume | Up to 10 min of head up tilt
  The primary outcome will be the percent change from supine in stroke volume during HUT

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Autonomic Dysfunction Center/ Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No